CLINICAL TRIAL: NCT04252157
Title: The Effect of Kinesiotaping on Saliva Control in Children With Cerebral Palsy
Brief Title: Taping for Saliva Control in Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, aydan aytar, assoc. prof., Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA 19/316
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy
Keywords: saliva; taping
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- kinesiotaping (Experimental): Kinesotape will be apply with suitable tension and necessery region.
  Interventions: Other: Kinesiotaping
- plesebo taping (Placebo Comparator): Tape will be appy with randomly region without tension.
  Interventions: Other: Plesebo Taping
- control (Other): Nothing will be applied
  Interventions: Other: Control

INTERVENTIONS:
Other: Kinesiotaping — Kinesiotape will be applied to the group. During the orbicularis oris muscle, I tape will be applied around the lip with a mechanical correction technique with 50-75% tension. I tape will be applied just below the Hyoid with a 50-75% tension mechanical correlation technique.
  Arms: kinesiotaping
Other: Plesebo Taping — An approximately 5 cm I tape will be applied to the group without applying any tension to the temporomandibular attachment for placebo taping.
  Arms: plesebo taping
Other: Control — no kinesio or tape will be applied
  Arms: control

SUMMARY:
This study aim to investigate the effect of banding on saliva control and quality of life in children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy describes a whole set of permanent disorders or disorders in the development of movement and posture, attributed to non-progressive disorders occurring in the developing fetal or infant brain, causing activity limitation. Motor disorders are often accompanied by sensory, perception, communication and behavioral disorders, epilepsy and secondary musculoskeletal problems.

Kinesio Taping has been proven to increase local circulation, reduce local edema and provide a positional stimulus for muscle, skin, or facial structures, regulating sensory input, and activating regions in the brain. KT is currently used to improve oral control in children with neurological and neuromuscular disorders and provides a reduction in saliva flow and frequency. However, knowledge of the potential of using neuromuscular bandages to manage the dribble flow has been limited.

ELIGIBILITY:
Inclusion Criteria:

* Being a dribble control disorder,
* Having a diagnosis of cerebral palsy,
* Being between the ages of 5-15,
* Not allergic to Kinesio Taping tape.

Exclusion Criteria:

* Using drugs for saliva control disorder,
* Botulinum toxin has been applied in the last 6 months,
* Active infection (tooth, intestine, etc.),
* Failure to comply with treatment,
* Swallowing disorder.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2021-03-17 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic Features | baseline
  Sociodemographic information such as age, gender, height, weight, education level of the parents will be asked.
Saliva Flow Amount | 2 days after taping
  The drool flow rate of children will be evaluated with DQ5m ("Drooling Quotient 5 minute"). Saliva flow rate can be evaluated by a standard observation of 5 minutes. The test is applied at least 1 hour after eating. Two separate measurements are taken in resting position, at rest and during any activity. The mouth must be empty and clean before the evaluation begins and if there is a saliva it will be removed. The evaluation is done every 15 seconds for 5 minutes and 1 point is given if there is a drooping out of the jaw and / or clothing. If there is no saliva output within 15 seconds, 0 is given. The evaluation is completed in 20 periods. When these periods are completed after 5 minutes, the data obtained are calculated with the formula. The result obtained is interpreted (0 = no new saliva flow 100% = new saliva flow in all periods). The application is valid and reliable.
Intensity and Frequency of Dribble Flow | 2 days after taping
  The "Saliva Severity and Frequency Scale" will be used to measure the severity and frequency of children's drool flow. Scale dribble intensity 0- No dribble 1- Light dribble (Only wet lips) 2- Moderate dribble (Drip on wet lips and chin) 3- Dribble dribble (Dribble drops to chin, from there to clothes) 4- Too much dribble (Dribble to clothes and objects drips) as a 0-4 score. It ranks the saliva frequency from 0 to 3 as follows; 0. No dribble 1. Rare dribble 2. Frequent dribble 3. Constant flowing dribble. The scale is valid and reliable.

SECONDARY OUTCOMES:
Posture Evaluation | 2 days after taping
  Posture evaluation will be done observationally. In this evaluation, anterior, posterior and lateral head, neck, and trunk posture will be evaluated.
Evaluation of the Effect on Family | 2 days after taping
  "Family Impact Scale" will be used to evaluate the effect of drool control disorder in children on the family. The scale, which consists of financial burden, familial and social impact, personal strain and coping sub parameters, is applied by answering the judgments about these parameters, fully agree, disagree and disagree at all. According to the total score received, comments are made about the level of influence of the family. A minimum score of 24 and a maximum of 96 can be obtained from the scale. The items in the scale are generally related to social, financial and emotional areas, and the high scale score indicates that the problem of mothers is high.The test is valid and reliable.
The Gross Motor Function Classification System Assesment | 2 days after taping
  The Gross Motor Function Classification System Assesment will be used to determine the level of cerebral palsy on the basis of self-initiated movement abilities.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided